CLINICAL TRIAL: NCT04449575
Title: Hand Eczema in the Health Care Sector
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: Statens Serum Institut (Other)
Responsible Party: Principal Investigator, Yasemin Topal Yüksel, MD, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: H20007169
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Hand Eczema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Bacteria from the skin will be sampled by eSwabs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health care workers with hand eczema: Swabs will be taken from eczema lesions on dominating hand (if possible) and nostril
  Interventions: Other: eSwabs
- controls (health care workers without hand eczema): swabs will be taken from healthy skin on dominating hand and nostril
  Interventions: Other: eSwabs

INTERVENTIONS:
Other: eSwabs — from skin

SUMMARY:
This project aims to investigate the prevalence of bacterial colonization and associated factors in health care workers with hand eczema with focus on Staphylococcus aureus.

DETAILED DESCRIPTION:
Two groups will be examined in this study: health care workers with HE and matched controls invited through a questionnaire study which will be sent to approximately 4000 health care workers in Capital Region. Samples from health care workers with and without hand eczema will be collected after obtaining their written informed consent. Collection of samples: Swabs will be rubbed on the skin for 30 seconds on lesional and non-lesional skin on the dominating hand and from the nostrils. The swabs will immediately be stored in -80 C° (research biobank) for subsequent analysis at Statens Serum Institute.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of hand eczema (for group with hand eczema)

Exclusion Criteria:

* Other skin diseases (in both groups)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health care workers from 4 hospitals in Capital Region, Denmark, with and without hand eczema.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Staphyloccous aureus presence | Baseline, cross-sectional
  Prevalence of S. aureus colonization on hands and in nose in two groups of health care workers. The swab samples will be assessed by culturing on selective S. aureus plates (chromID S. aureus; bioMerieux, Marcy l'Etoile, France) and incubated overnight at 37 °C. DNA will be purified from S. aureus isolates using the Qiagen DNeasy Blood and Tissue Purification Kit (Qiagen, Hilden, Germany).

SECONDARY OUTCOMES:
CC-types and spa-typing | Baseline, cross-sectional
  clonal complex (CC) type and spa-types are characterizing the S. aureus. Will be correlated to departments and professions of health care workers. The S. aureus will be further characterized by spa typing, which will be performed by polymerase chain reaction and Sanger sequencing of the product. The respective CC types will be assigned from the spa type using eBURST (http://eburst.mlst.net).
Hand Eczema Severity Index (HECSI) | Baseline, cross-sectional
  Validated severity measurement tool for hand eczema performed by the investigator. Severity will be correlated to S. aureus colonization and CC types

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin T. Yüksel, MD, Principal Investigator — University of Copenhagen Bispebjerg and Frederiksberg Hospital; Tove Agner, MD, PhD, Study Director — University of Copenhagen Bispebjerg and Frederiksberg Hospital
Locations (1):
- Yasemin Topal Yüksel, Copenhagen, KBH NV, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mernelius S, Carlsson E, Henricson J, Lofgren S, Lindgren PE, Ehricht R, Monecke S, Matussek A, Anderson CD. Staphylococcus aureus colonization related to severity of hand eczema. Eur J Clin Microbiol Infect Dis. 2016 Aug;35(8):1355-61. doi: 10.1007/s10096-016-2672-2. Epub 2016 May 19. PMID 27193891
- [Background] Haslund P, Bangsgaard N, Jarlov JO, Skov L, Skov R, Agner T. Staphylococcus aureus and hand eczema severity. Br J Dermatol. 2009 Oct;161(4):772-7. doi: 10.1111/j.1365-2133.2009.09353.x. Epub 2009 Jul 3. PMID 19575755
- [Background] Pittet D, Allegranzi B, Sax H, Dharan S, Pessoa-Silva CL, Donaldson L, Boyce JM; WHO Global Patient Safety Challenge, World Alliance for Patient Safety. Evidence-based model for hand transmission during patient care and the role of improved practices. Lancet Infect Dis. 2006 Oct;6(10):641-52. doi: 10.1016/S1473-3099(06)70600-4. PMID 17008173
- [Background] Brans R, Kolomanski K, Mentzel F, Vollmer U, Kaup O, John SM. Colonisation with methicillin-resistant Staphylococcus aureus and associated factors among nurses with occupational skin diseases. Occup Environ Med. 2016 Oct;73(10):670-5. doi: 10.1136/oemed-2016-103632. Epub 2016 Jun 29. PMID 27358469
- [Background] Clausen ML, Edslev SM, Norreslet LB, Sorensen JA, Andersen PS, Agner T. Temporal variation of Staphylococcus aureus clonal complexes in atopic dermatitis: a follow-up study. Br J Dermatol. 2019 Jan;180(1):181-186. doi: 10.1111/bjd.17033. Epub 2018 Oct 10. PMID 30070683
- [Background] Held E, Skoet R, Johansen JD, Agner T. The hand eczema severity index (HECSI): a scoring system for clinical assessment of hand eczema. A study of inter- and intraobserver reliability. Br J Dermatol. 2005 Feb;152(2):302-7. doi: 10.1111/j.1365-2133.2004.06305.x. PMID 15727643